CLINICAL TRIAL: NCT01337622
Title: Gastric Residuals in Preterm Infants (GRIP)
Brief Title: Gastric Residuals in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster Children's Hospital (Other)
Responsible Party: Principal Investigator, Christoph Fusch, Division head NICU, McMaster Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201101GRIP
Record Dates: First submitted 2011-04-15; First posted 2011-04-19 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Early Enteral Feeding Advancement; Nutrition; Preterm Infants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No routine check for gastric residuals (Experimental)
  Interventions: Procedure: No check of gastric residuals for early enteral feeding advancement
- Routine check for gastric residuals (Active Comparator)
  Interventions: Procedure: Routine check of gastric residuals for early enteral feeding advancement

INTERVENTIONS:
Procedure: No check of gastric residuals for early enteral feeding advancement — Discontinuation of gastric feeding and its advancement will be based on clinical examination of the abdomen and gastric aspirates containing blood or significant vomiting.
  Arms: No routine check for gastric residuals
Procedure: Routine check of gastric residuals for early enteral feeding advancement — Discontinuation of gastric feeding and its advancement will be based on current practice of clinical examination of the abdomen and checking residual before every feed. Volume and color of gastric residual will be considered according to the current guideline.
  Arms: Routine check for gastric residuals

SUMMARY:
Checking of gastric residuals prior to the continuation/increase of enteral feeding prolongs the time to establish full gastric feeding in the early postnatal period.

ELIGIBILITY:
Inclusion Criteria:

* Infants with a birth weight ≥ 1500g and < 2000g
* Age ≤48 hours of life
* Informed, written parental consent

Exclusion Criteria:

* Antenatally recognized gastrointestinal malformation
* Major congenital anomaly
* Chromosomal anomaly
* NEC stage II
* Severe acidosis, asphyxia (pH <7.0)
* Severe growth restriction below 3rd percentile

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Time to reach full enteral feeding | from inclusion (during first 48h of life) until 1 month
  Full enteral feeding is defned as an milk intake of equal or more than 120 ml/kg/d.

SECONDARY OUTCOMES:
growth, tolerance, morbidity | from inclusion (during first 48h of life) until one month
  Time to regain birth weight and maintain weight gain. Incidence of sepsis from birth until 48 hours after parenteral nutrition was administered.
  Use of antibiotics. Incidence of feeding intolerance and necrotizing enterocolitis.

CONTACTS AND LOCATIONS:
Overall Officials: Sumesh Thomas, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Singh B, Rochow N, Chessell L, Wilson J, Cunningham K, Fusch C, Dutta S, Thomas S. Gastric Residual Volume in Feeding Advancement in Preterm Infants (GRIP Study): A Randomized Trial. J Pediatr. 2018 Sep;200:79-83.e1. doi: 10.1016/j.jpeds.2018.04.072. Epub 2018 Jun 1. PMID 29866595